CLINICAL TRIAL: NCT05822388
Title: A Neural Basis for Cognitive Decline Following Deep Brain Stimulation
Brief Title: Cognitive Decline Following Deep Brain Stimulation
Status: Recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00125181
Record Dates: First submitted 2023-04-10; First posted 2023-04-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson's Disease undergoing DBS: This study will recruit 55 patients with Parkinson's disease (PD) participants who will undergo DBS surgery and and are scheduled for a pre-DBS neuropsychological evaluation at MUSC.
  Interventions: Procedure: Deep Brain Stimulation Surgical Procedures as Part of Routine Clinical Care
- Healthy Control participants without Parkinson's Disease: This study will recruit 25 healthy controls (age-matched) to serve as a comparison of baseline cognitive and neuroimaging measures.

INTERVENTIONS:
Procedure: Deep Brain Stimulation Surgical Procedures as Part of Routine Clinical Care — Participants in this study will already be undergoing a DBS intervention, however, this is part of their standard clinical care. Pre-surgical DBS candidates that enroll in this study will consent to participate in 1) pre-operative neuroimaging including a high-resolution MRI scan, 2) collection of pre-operative neurocognitive data via chart review and 3) a 1-year postoperative neurocognitive assessment.
  Groups: Parkinson's Disease undergoing DBS

SUMMARY:
This research study aims to identify MRI-based brain biomarkers that predict an individual's response to Deep Brain Stimulation (DBS). In particular, this study will focus on changes in cognition associated with DBS. A total of 55 participants with Parkinson's Disease planning to undergo DBS will be recruited from MUSCs Clinical DBS Program. Participants will undergo four visits, including a 1-hour screening visit, a 1.5-hour pre-DBS MRI scanning visit, and a 3.5-hour post-DBS cognitive assessment visit. In addition control participants without Parkinson's Disease will be recruited to undergo MRI scanning and cognitive assessments.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) targeting the subthalamic nucleus (STN) is a well-established surgical intervention to treat Parkinson's Disease (PD) patients with disabling motor fluctuations and dyskinesias. Although this therapy is effective for motor complications, a subset of patients will go on to experience cognitive decline, which can overshadow improvements in the quality of life provided by STN-DBS. This accelerated decline in cognition occurs in patients despite rigorous evaluation of their neuropsychological status prior to surgery. While the factors contributing to cognitive decline following DBS remain unclear, there is evidence this may be the result of 1) limited cognitive reserve prior to DBS surgery, 2) stimulation that interferes with cognitive networks, and/or 3) a microlesion effect due to placement of the lead. Understanding how these factors contribute to DBS-induced cognitive decline has the potential to improve patient selection for surgery and optimize the selection of stimulation targets that minimize undesirable cognitive side effects.

ELIGIBILITY:
PD Participants

Inclusion Criteria:

* Subjects above 18 years of age
* Subjects who will undergo DBS surgery as part of their clinical care for PD

Exclusion Criteria:

* Uncorrected visual or hearing impairments, as indicated by self-report
* Individuals who are pregnant or expect to become pregnant during the course of the study
* Individuals with claustrophobia, or the inability to lie supine position in the MRI scanner
* COPD with oxygen dependence
* Non-MRI compatible metal implants (surgical clips or staples, cardiac pacemakers etc.)

Non-PD Control Participants

Inclusion Criteria:

* Subjects above 18 years of age
* Age matched to participants in PD group

Exclusion Criteria:

* Diagnosis of Parkinsons Disease or other movement disorder
* Untreated neuropsychiatric disorders
* Uncorrected visual or hearing impairments, as indicated by self-report
* Individuals who are pregnant or expect to become pregnant during the course of the study
* Individuals with claustrophobia, or the inability to lie supine position in the MRI scanner
* COPD with oxygen dependence
* Non-MRI compatible metal implants (surgical clips or staples, cardiac pacemakers etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease (PD) participants who will undergo DBS surgery and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition | From the DBS candidacy evaluation stage (approximately one month prior to deep brain stimulation) until 1 year post surgery
  Change in cognitive performance using a comprehensive neuropsychological battery (e.g., language, executive control, memory, and attention)
Brain Microstructure (DKI) | Within the DBS candidacy evaluation stage (approximately one month prior to deep brain stimulation (DBS))
  Nucleus Basalis of Meynert (NBM) and striatal microstructural integrity using diffusion kurtosis imaging (mean kurtosis; MK)

SECONDARY OUTCOMES:
Brain Functional Connectivity | Within the DBS candidacy evaluation stage (approximately one month prior to deep brain stimulation (DBS))
  Functional connectivity in cognitive networks including the Nucleus Basalis of Meynert (NBM) and the striatum
Brain Microstructure (DTI) | Within the DBS candidacy evaluation stage (approximately one month prior to deep brain stimulation (DBS))
  Nucleus Basalis of Meynert (NBM) and striatal microstructural integrity using diffusion tensor imaging (mean diffusivity; MD)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Lench, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No